CLINICAL TRIAL: NCT04467437
Title: Transcutaneous Spinal Stimulation With Intensive Gait Training for Individuals With Neurologic Conditions
Brief Title: Transcutaneous Stimulation for Neurological Populations
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Chet Moritz, Associate Professor of Electrical & Computer Engineering and Rehabilitation Medicine, University of Washington
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00008896
Record Dates: First submitted 2020-07-07; First posted 2020-07-13 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Neurological Disorder; Cerebral Palsy
Keywords: Spinal Electrical Stimulation; Treadmill Training
MeSH Terms: conditions — Nervous System Diseases; Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intensive Training Only (Active Comparator): Physical and gait training that targets rehabilitation of walking function.
  Interventions: Other: Gait Training
- Intensive Training Combined with Spinal Stimulation (Active Comparator): Transcutaneous spinal stimulation combined with physical and gait training that targets rehabilitation of walking function.
  Interventions: Other: Gait Training; Device: Transcutaneous Spinal Stimulation

INTERVENTIONS:
Other: Gait Training — Training that targets rehabilitation of walking function
Device: Transcutaneous Spinal Stimulation — Non-invasive electrical stimulation of the spinal cord over the skin combined with gait training
  Arms: Intensive Training Combined with Spinal Stimulation

SUMMARY:
The purpose of the study is to evaluate whether non-invasive stimulation over the spinal cord at the neck and/or lower back can improve walking function for people with neurologic conditions. Spinal stimulation has been used extensively for individuals with spinal cord injury, and has demonstrated improvements in function. This study will extend this work to other neurologic conditions, such as cerebral palsy and stroke, that also demonstrate similar impairments as spinal cord injury.

The primary aims of this study are to:

Aim 1: Evaluate impact of spinal stimulation on spasticity and locomotor function.

Aim 2: Investigate participant perceptions of spinal stimulation.

The investigators will be using a cross-over design study to compare intensive training only to intensive training combined with spinal stimulation. After an initial baseline period of up to 4 weeks (Phase I). Participants will have their first intervention phase of the study (Phase II). This will involve either intensive training only (Condition A) or intensive training combined with spinal stimulation (Condition B). This will be followed by a washout period with no intervention (Phase III) and then the second intervention phase (Phase IV). The second intervention phase will involve either Condition A or Condition B, whichever the participants did not received during Phase II. Phases II-IV will each last up to 8 weeks. After the intervention period is complete, the participant will be asked to come for follow-up visits up to 3 months after the intervention phases are completed (Phase V).

ELIGIBILITY:
Inclusion Criteria:

* have a neurologic condition
* can walk 20 yards, with or without an assistive device
* have stable medical condition
* are capable of performing simple cued motor tasks and who can follow 2-3 step commands
* have ability to attend up to 5 sessions per week physical therapy sessions and testing activities
* have adequate social support to be able to participate in training and assessment sessions, up to 5 sessions per week, for the duration of up to 11 months within the study period.
* who are volunteering to be involved in this study
* can read and speak English

Exclusion Criteria:

* have significant medical disease; including uncontrolled systemic hypertension with values above 170/100 mmHg; cardiac or pulmonary disease; uncorrected coagulation abnormalities or need for therapeutic anticoagulation.
* have cardiovascular or musculoskeletal disease or injury that would prevent full participation in physical therapy intervention
* have a history of uncontrolled seizures
* have unhealed fracture or other musculoskeletal impairment that might interfere with lower extremity rehabilitation or testing activities
* are dependent on ventilation support
* have implanted stimulator (e.g. epidural stimulator, vagus nerve stimulator, pacemaker, cochlear implant, etc) or drug delivery device (e.g. baclofen pump)
* have history of orthopedic surgery in lower extremities or neurosurgery that may be a confounding factor for interpretation of the results (such as tendon transfer, tendon or muscle lengthening for spasticity management, injection therapies to lower extremity muscles, etc.) in last 12 months
* have established osteoporosis and taking medication for osteoporosis treatment.
* have rheumatic diseases (rheumatoid arthritis, systemic lupus erythematosus, etc.)
* have active cancer

Ages: 4 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline - Six Minute Walk Test | Measurements at baseline and repeated measurements once every two weeks throughout the study, an average of 10 months.
  Measure of walking ability. The distance is reported in meters.
Change from baseline - Ten Meter Walk Test | Measurements at baseline and repeated measurements once every two weeks throughout the study, an average of 10 months.
  The measure of walking ability at fast and self-selected speeds. The walking speed is reported as meters per second.

SECONDARY OUTCOMES:
Change from baseline - Kinetic and kinematic gait analysis using three dimensional camera system | Measurements at baseline and repeated measurements once every two months throughout the study, an average of 10 months.
  Measurement of leg function and walking ability. Joint angle is reported in angle degrees, and velocity is reported in meters per second. Kinematic analysis will able to used to measure gait coordination and spatiotemporal outcomes, such as step length and step time.
Change from baseline - Electromyography recording of lower extremity muscles | Measurements at baseline and repeated measurements once every two months throughout the study, an average of 10 months.
  Measurement of muscle and nerve functions. The muscle activities are reported in micro-volts.
Change from baseline - Gait Outcomes Assessment List | Measurements at baseline and repeated measurements once every two months throughout the study, an average of 10 months.
  The patient-reported outcome measure for ambulatory children with cerebral palsy. The Gait Outcomes Assessment List comprises 48 items distributed across 7 subscales and spans all domains of the International Classification of Functioning, Disability, and Health. The score range is between 0 and 100. The higher scores mean a better outcome.
Change from baseline - Timed Up and Go | Measurements at baseline and repeated measurements once every two months throughout the study, an average of 10 months.
  Measurement of mobility and fall risk. The time to complete the test is recorded in seconds.
Change from baseline - Modified Ashworth and Tardieu Scales | Measurements at baseline and repeated measurements once every two weeks throughout the study, an average of 10 months.
  Measurement of spasticity in muscles. The score range is between 0 and 5. The lower scores mean a better outcome.
Change from baseline - Patient-Reported Outcomes Measurement Information System Pediatric Profile | Measurements at baseline and repeated measurements once every two months throughout the study, an average of 10 months.
  Includes six domains. These are depression, Anxiety, Physical Function-Mobility, Pain Interference, Fatigue, and Peer Relationships. Each domain contains 8 items, along with a single item on Pain Intensity scored between 0 to 10.
  The score range for each domain is between 1 and 5. The lower scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine M Steele, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No